CLINICAL TRIAL: NCT05010798
Title: Quality of Life in Binge Eating Disorder: Danish Language Disease Specific Measures.
Brief Title: Quality of Life in Binge Eating Disorder.
Status: Completed | Type: Observational
Sponsor: Odense University Hospital (Other)
Collaborators: University of Southern Denmark (Other); Region of Southern Denmark (Other)
Responsible Party: Principal Investigator, René Klinkby Støving, Professor, Odense University Hospital
Other Study IDs: QoL BED
Record Dates: First submitted 2021-08-10; First posted 2021-08-18 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Binge-Eating Disorder; Quality of Life
Keywords: binge eating disorders; Quality of life
MeSH Terms: conditions — Binge-Eating Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Binge Eating Disorder (BED) patients tend to report low quality of life (Qol). However, research is limited. Most research on Qol in BED include generic measures, rather than disease specific. Obesity is prevalent in BED, but contradicting evidence exists on the influence of obesity in BED.

DETAILED DESCRIPTION:
Eating disorders (ED's) are a group of disorders characterized by abnormal eating behaviors ranging from insufficient to excessive food intake, with concurrent disturbances in thoughts and emotions. Binge Eating Disorder (BED) is the most prevalent ED in both men and women, yet was only recently included in the Diagnostic and Statistical Manual of Mental Disorders fifth edition (DSM-5) as a diagnostic entity.

In general, ED's have been associated with significantly worse health related quality of life (HRQoL) compared to healthy population.

High rates of overweight (BMI ≥ 25) and obesity (BMI ≥ 30) are found in BED patients and obesity in itself is associated with lower QoL. The most widely used tools to measure Qol in ED's are the Medical Outcome Studies Short Form (SF) Scale, e.g. SF-36 and SF-12, which are generic in nature. Generic QoL measures have shown lack of sensitivity for some ED diagnoses and might not be suitable enough to pick up unique features that might characterize each disorder.

The objective of this study is to evaluate quality of life in Danish BED patients before treatment by using disease specific Qol measure. Furthermore, we want to assess the impact of obesity and depression on disease specific Qol in BED patients. The hypothesis are that obesity and depression will be associated with an impaired level of disease specific Qol.

ELIGIBILITY:
Inclusion Criteria:

1. Patients referred to treatment for BED at Center f. Eating Disorders, OUH.

Exclusion Criteria:

1. Extremely severe BED.
2. Severe psychiatric comorbidity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred to treatment for BED at Center f. Eating Disorders, OUH. This is a new and free treatment offer. The population is therefore not known in advance, but is expected to be quite heterogeneous.
Sampling Method: Non-Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
Eating Disorder Quality of Life Questionnaire (EDQLS) | Approximately 2 years
  Disease specific quality of life measure.
  The EDQLS consists of 40 items across 12 subscales and takes 2-11 minutes (mean 5 minutes) to complete. Each item is rated on a five-point Likert scale from 'strongly disagree' (scored as 1) to 'strongly agree' (scored as 5), with a higher score indicating better HRQoL (minimum score 40; maximum score 200).
  The 12 subscales are: cognitive, education/vocation, family and close relationships, relationships with others, future outlook, appearance, leisure, psychological, emotional, values and beliefs, physical, and eating. Each subscale contains three items, except for the 'eating' subscale which has six items. The EDQLS software includes an automatic scoring program that converts all item responses to a total score (some subscales require reverse scoring prior to summing).

CONTACTS AND LOCATIONS:
Overall Officials: René K Støving, PhD, Principal Investigator — Odense UH
Locations (2):
- Denmark (2):
  - Center for eating Disorders, Odense University Hospital, Odense
  - Department of Endocrinology, Odense University Hospital, Odense

REFERENCES:
- [Background] Winkler LA, Gudex C, Lichtenstein MB, Roder ME, Adair CE, Sjogren JM, Stoving RK. Explanatory Factors for Disease-Specific Health-Related Quality of Life in Women with Anorexia Nervosa. J Clin Med. 2021 Apr 9;10(8):1592. doi: 10.3390/jcm10081592. PMID 33918786
- [Derived] Gudmundsdottir S, Linnet J, Lichtenstein MB, Adair CE, Carlsson SD, Brandt L, Rasmussen J, Stoving RK. Low quality of life in binge eating disorder compared to healthy controls. Dan Med J. 2023 Mar 14;70(4):A07220443. PMID 36999814